CLINICAL TRIAL: NCT05421182
Title: Psychological Impact of Medical Evacuations on Families of Patients Admitted to Intensive Care Unit for Severe COVID-19
Acronym: IPES-CoV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHMS21004
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — COVID-19; Stress Disorders, Post-Traumatic | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Critical Care

STUDY DESIGN:
Intervention Model Description: Case-Control Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interview of the trusted person of evacuated patient (Other): The interview of the trusted person of evacuated patient will be done 8 months (+/-2 months) after the medical evacuation.
  The interview will be carried out by a psychologist or by a doctor from the ICU
  Interventions: Other: Revised Impact of Event Scale; Other: Hospital Anxiety and Depression scale; Other: 36-Item Short Form Survey; Other: satisfaction survey; Other: semi-directed interview with trusted person on the general experience of the patient's medical evacuation
- Interview of the trusted person of the not evacuated patient (Other): The interview of the trusted person of the not evacuated patient will be done 8 months (+/-2months) after the ICU admission The interview will be carried out by a psychologist or by a doctor from the ICU.
  Interventions: Other: Revised Impact of Event Scale; Other: Hospital Anxiety and Depression scale; Other: 36-Item Short Form Survey; Other: satisfaction survey; Other: semi-directed interview with trusted person on the general experience of hospitalization in intensive care

INTERVENTIONS:
Other: Revised Impact of Event Scale — to measure the affect of routine life stress,everyday traumas and acute stress
  Other Names: IES-R
Other: Hospital Anxiety and Depression scale — to measure anxiety and depression
  Other Names: HADS
Other: 36-Item Short Form Survey — SF-36 is a set of generic, coherent, and easily administered quality-of-life measures.
  Other Names: SF-36
Other: satisfaction survey — satisfaction survey of the trusted person about the communication with ICU personal
Other: semi-directed interview with trusted person on the general experience of the patient's medical evacuation — interview of the trusted person about the medical evacuation : evacuation announcement;organization of the medical evacuation,; concerns related to evacuations;reception and information by the center admitting the evacuated patient; arrangements of visit, patient repatriated
  Arms: Interview of the trusted person of evacuated patient
Other: semi-directed interview with trusted person on the general experience of hospitalization in intensive care — interview of the trusted person about ICU hospitalization: reception in ICU; ICU organization; concerns related to ICU hospitalization, information and communication with ICU staff, arrangements of visit, context of ICU discharge
  Arms: Interview of the trusted person of the not evacuated patient

SUMMARY:
At the "Métropole Savoie" hospital, to deal with the daily influx of severe patients during the second wave of COVID-19, 23 patients had to be transferred away from their home city and far from their families as part of a medical evacuation (EVASAN).

The purpose of the study is to investigate whether there is an association between medical evacuations and the occurrence of psychological disorders such as post-traumatic stress, anxiety or depression occurring within 6 to 10 months in families of evacuated patients.

The investigators want to compare the prevalence of psychological disorders in the families of patients evacuated for a serious form of COVID-19 (cases) compared to that of families of patients not evacuated (controls) hospitalized for a serious form of COVID-19.

DETAILED DESCRIPTION:
The case group is trusted person of evacuated patient. The control group is trusted person of not evacuated patient.

The trusted person of the group control will be matched to trusted patient of the case group on :

their relationship with the patient (spouse/ascendant/descendant/other) and on criteria specific to the patient: sex, age range ( <75 years or ≥ 75 years), invasive ventilation and becoming at 3 months post COVID-19 (survivor / non survivor)

ELIGIBILITY:
Inclusion Criteria:

Trusted person of patients admitted to the Adult Intensive Care Unit (ICU) of the "Metropole Savoie"hospital

* during the second wave of COVID-19 in France
* for a serious form of COVID-19
* hospitalized more than 72 hours in ICU

the case group is trusted person of evacuated patient. the control group is trusted person of not evacuated patient.

Non -inclusion criteria :

Trusted Person Refusing patient Medical Evacuation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the prevalence of post-traumatic stress disorder, among families of patients with severe COVID-19 evacuated to another region (case) compared to families of matched patients with severe COVID-19 not evacuated to another region (controls). | at 8months (+/-2 months) after medical evacuations for the case group, and at 8 months (+/-2 months) after ICU admission for the control group
  the post-traumatic stress disorder of the trusted person is assessed by the Impact of Event Scale - Revised (IES-R), at 8months (+/-2 months) after medical evacuations for the case group, and at 8 months (+/-2 months) after Intensive Care Unit (ICU) admission for the control group

SECONDARY OUTCOMES:
Prevalence of anxiety and/or depression symptoms questionnaire in families of patients hospitalized with severe COVID-19. | at 8 months (+/- 2months) in families of patients hospitalized in intensive care for a serious form of COVID-19.
  Association between medical evacuations and the occurrence of symptoms of anxiety and/or depression at 8 months in families of patients hospitalized in intensive care for a serious form of COVID19. anxiety and/or depression symptoms assessed by the Hospital Anxiety and Depresion Scale (HADS)
Quality of Life in families of patients with severe COVID-19 | at 8 months (+/- 2months) in families of patients hospitalized in intensive care for a serious form of COVID-19.
  Quality of Life assessed by Medical Outcomes Study Short Form 36 (SF-36)
Satisfaction with the communication between the health care team and the family of the patient hospitalized with severe form of COVID19 | at 8 months (+/- 2months) in families of patients hospitalized in intensive care for a serious form of COVID-19.
  satisfaction is measured using a simple digital scale,
Qualitative analysis by a psychologist of a semi-structured interview of the testimony and specific experience of families at 8 months. | at 8 months (+/- 2months) in families of patients hospitalized in intensive care for a serious form of COVID-19.
  semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Peigne, Principal Investigator — CH Metropole Savoie
Locations (1):
- CH Metropole Savoie, Chambéry, France

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study, will not be available to other researchers